CLINICAL TRIAL: NCT01774747
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Oral Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of DSP-1053 in Healthy Subjects and in Subjects With Major Depressive Disorder
Brief Title: A Multiple Ascending Oral Dose Evaluation of the Safety, Tolerability, and Pharmacokinetics of DSP-1053 and Its Metabolites in Healthy Subjects and in Subjects With Major Depressive Disorder
Acronym: MAD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This program was terminated for financial reasons
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7750090
Record Dates: First submitted 2013-01-08; First posted 2013-01-24 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DSP-1053 (Experimental): DSP-1053 10, 15, 20, 30, 45, 60, 90 mg once daily for 14 days
  Interventions: Drug: DSP-1053; Drug: Placebo
- Placebo (Placebo Comparator): Placebo 10, 15, 20, 30, 45, 60, 90 mg once daily for 14 days
  Interventions: Drug: DSP-1053; Drug: Placebo

INTERVENTIONS:
Drug: DSP-1053 — DSP-1053 10, 15, 20, 30, 45, 60, 90 mg once daily for 14 days
Drug: Placebo — Placebo 10, 15, 20, 30, 45, 60, 90 mg once daily for 14 days

SUMMARY:
Double-blind, placebo-controlled, multiple ascending oral dose evaluation of the safety, tolerability, and pharmacokinetics of DSP 1053 and its metabolites in healthy subjects and in subjects with major depressive disorder

DETAILED DESCRIPTION:
This study will be conducted at a single site as a double-blind, placebo-controlled, mulitple ascending oral doses evaluation of the safety, tolerability, and pharmacokinetics of DSP-1053 and its metabolites in healthy subjects with Major depressive disorder after the minimumally intolerated dose is reached in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects:

Be able to understand and willing to sign the Informed Consent Form, and capable of providing written authorization for use and disclosure of protected health information per requirements of 45 Code of Federal Regulations (CFR) 164.508 (Health Information Portability and Accountability Act [HIPAA]).

Be healthy male or female subjects between 18 and 50 years of age (inclusive). Have a BMI 18 and 33 kg/m2. Have no clinically relevant abnormal laboratory values at screening and Day -1.

Have no clinically relevant findings from vital sign measurements at screening and check-in.

Have no clinically relevant findings from physical examination at screening and check in.

Have a negative urine drug of abuse test (cannabinoids, barbiturates, cocaine, opiates, benzodiazepines, phencyclidine, and methadone) and negative cotinine test at screening and check in.

Have a negative alcohol breath test at screening and check in. Have a negative Hepatitis B surface antigen, Hepatitis C antibody, and human immunodeficiency virus (HIV) antibody tests at screening.

Have normal hepatic function [aspartate transaminase (AST), bilirubin, and alanine transaminase (ALT)] and renal function (creatinine clearance greater than 80 mL/min as assessed by Cockcroft Gault equation using serum creatinine) at screening and Day 1.

Be females who are of childbearing potential:

have a negative serum hCG pregnancy test at screening and Day -1; willing to not breastfeed from Day -5 until 90 days after discharge from the study site;

Be females who are:

unable to have children (eg, post menopausal, tubal ligation, hysterectomy) OR willing to remain abstinent (not engage in sexual intercourse) from check in until 90 days after discharge from the study site.

OR willing to use an effective method of double-barrier birth control (eg, partner using condom and female using diaphragm, contraceptive sponge, spermicide, or intrauterine device) from check-in until 90 days after discharge from the study site.

Be males who:

are sterile or willing to remain sexually abstinent or use an effective method of birth control (eg, condom) from check-in until 90 days after discharge from the study site.

AND agree not to donate sperm during the study and for 90 days after discharge from the study site.

Refrain from strenuous physical activity from 48 hours prior to check-in until discharge from the study site.

Agree to remain housed at the study site for the clinical confinement of study and return for any visits required for additional safety or PK assessments.

Agree to consume study meals per protocol.

Subjects with MDD:

In addition to inclusion criteria mentioned above for healthy subjects, the following inclusion criteria will be applied to subjects with MDD:

Have the diagnosis of MDD as defined by the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition; Text Revision (DSM IV TR) criteria and confirmed by the Mini International Neuropsychiatric Interview (MINI) diagnostic interview. This diagnosis will be confirmed by a psychiatrist or psychologist. The diagnosis should be supplemented (when possible) by confirmation of chart records or by a discussion with a treating healthcare professional or reliable informant. Diagnosis made by a psychologist must be reviewed by a psychiatrist.

The subjects' current major depressive episode must be ≥ 4 weeks and < 2 years in duration.

Are able to wash-out from prior antidepressant therapies by Day -1, are able to forego psychotherapy from Day -1 through Day 10, inclusive, and are deemed clinically stable by PI's assessment.

May have a comorbid anxiety disorder such as generalized anxiety disorder (GAD) or social phobia but not obsessive compulsive disorder (OCD) as long as the comorbid anxiety disorder is not the major source of impairment.

Have a stable living arrangement for at least 3 months prior to check in and agree to return to a similar living arrangement after discharge. This criterion is not meant to exclude subjects who have temporarily left a stable living environment. Such subjects remain eligible to participate in this study. Chronically homeless subjects should not be enrolled. The Medical Monitor should be consulted for individual cases as needed.

Exclusion Criteria:

Healthy Subjects

Significant history or clinical manifestations of any acute or chronic condition that in the opinion of the PI, would limit the subject's ability to complete and/or participate in the study:

metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders; drug hypersensitivity; stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (appendectomy, hernia repair, and/or cholecystectomy will be allowed at the discretion of the PI); abnormal ECG, which, in the PI's opinion, is clinically significant; known or suspected alcohol or substance abuse/ dependence within one year prior to check in; movement disorders including tremor; lifetime or family history of seizures or a febrile seizure. Poor peripheral venous access. Does not tolerate venipuncture. Donation of blood from 28 days prior to screening through study completion, inclusive.

Receipt of blood products within 2 months prior to check in. Any acute or chronic condition that, in the opinion of the PI, would limit the subject's ability to complete and/or participate in this clinical study.

Female subjects with menstrual dysfunction. Considered by the PI to be at imminent risk of suicide or injury to self, others, or property.

Subject answers "yes" to "Suicidal Ideation" Items 4 or 5 on the CSSRS at screening.

Subjects who, by history, have smoked or used tobacco products within 60 days from screening until study follow up.

Consumption of food or beverages containing alcohol, grapefruit, or caffeine within 72 hours prior to check in and until discharge from the study site, unless deemed acceptable by the PI.

Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half lives or 3 months prior to check-in, whichever is longer.

Taken any drug(s) known to be clinically relevant cytochrome P450 2D6 (CYP2D6), or cytochrome P450 3A4 (CYP3A4) inhibitors or inducers within 28 days prior to the first DSP 1053 dose and during the study conduct through follow up.

Taken any antihistamines within 14 days prior to check-in and during the study. Family history of prolonged QT interval (QTc) prolongation. Subjects, who by history, are at any risk for bleeding or have abnormal prothrombin values or currently use of anticoagulant treatment (such as warfarin) Clinically important folic acid or B12 abnormalities detected within 3 months before screening.

Use of any prescription medications/products within 14 days prior to check in unless deemed acceptable by the PI.

Subjects with MDD

Except for Exclusion Criterion 18 mentioned above for healthy subjects all exclusion criteria will be applied and in addition the following exclusion criteria will be applied to subjects with MDD:

History of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, eating disorder, or obsessive compulsive disorder.

Any current Axis I disorder other than major depressive disorder which is the focus of treatment.

Substance or alcohol abuse in the last 3 months or substance or alcohol dependence in the last 12 months.

Concomitant psychotropic medication, including herbals. Significant risk of violent behavior or a significant risk of suicidal behavior based on history or in the PI's judgment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To reach minimumally intolerable dose based on stopping criteria | 14 days
  * At least 50% of subjects within a cohort at dose level experience multiple moderate drug related adverse events or one severe drug-related adverse event
  * one drug related serious adverse event within a cohort at dose level
  * seizure of any severity or seriousness is observed in a subject who received DSP-1053
  * Mean plasma DSR_22898 Cmax greater or equal to 32ng/ml for a cohort

SECONDARY OUTCOMES:
Characterize the pharmacodynamic relationship based on serotonin transporter occupancy of DSP-1053 following multiple oral doses of DSP-1053 in healthy subjects and major depressive disorder subjects | 14 days
  Measurement of inhibition of active [H]-5HT transport in cells expressing the human serotonin transporter.
To characterize exposure of DSP-1053 and its metabolites (AUC, Cmax and Tmax) after multiple ascending dose of DSP-1053 | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, DSP-1053, Study Director — Sumitomo Pharma America, Inc.
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States